CLINICAL TRIAL: NCT00297479
Title: Group Therapy for Nicotine Dependence
Brief Title: Group Therapy for Nicotine Dependence: Mindfulness and Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2004-0988; R01DA018875 (NIH); NCI-2012-02081 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2006-02-24; First posted 2006-02-28 (Estimated); Results first posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Smoking; Tobacco Use Cessation
Keywords: Tobacco Cessation; Smoking Cessation
MeSH Terms: conditions — Smoking; Tobacco Use Cessation; Smoking Cessation | interventions — Therapeutics; Counseling; Nicotine; Psychotherapy, Group

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mindfulness-Based Treatment Group (MBAT) (Experimental): MBAT is 6 weeks of nicotine patch therapy; a Self-help guide; and In-person group therapy/counseling (8 sessions over 8 weeks) using a Mindfulness-Based Addiction Treatment for nicotine dependence.
  Interventions: Behavioral: MBAT Group Therapy; Drug: Nicotine
- Standard Care Group (Active Comparator): Standard Care Group (ST) is 6 weeks of nicotine patch therapy, a Self-help guide and In-person group therapy/counseling (8 sessions over 8 weeks) based upon Treating Tobacco Use and Dependence Clinical Practice Guideline
  Interventions: Drug: Nicotine; Behavioral: Group Therapy
- Usual Care Group (Active Comparator): Usual Care (UC) is 6 weeks of nicotine patch therapy, a Self-help guide and In-person individual counseling (4 sessions over 8 weeks) based upon Treating Tobacco Use and Dependence Clinical Practice Guideline
  Interventions: Drug: Nicotine; Behavioral: Individual Therapy

INTERVENTIONS:
Behavioral: MBAT Group Therapy — In-person group therapy/counseling (8 sessions over 8 weeks) using a Mindfulness-Based Addiction Treatment for nicotine dependence
  Other Names: therapy; counseling
  Arms: Mindfulness-Based Treatment Group (MBAT)
Drug: Nicotine — 6 weeks of nicotine patch therapy
  Other Names: nicotine patch therapy
Behavioral: Group Therapy — In-person group therapy/counseling (8 sessions over 8 weeks) based upon Treating Tobacco Use and Dependence Clinical Practice Guideline
  Other Names: counseling
  Arms: Standard Care Group
Behavioral: Individual Therapy — In-person individual counseling (4 sessions over 8 weeks) based upon Treating Tobacco Use and Dependence Clinical Practice Guideline
  Other Names: counseling
  Arms: Usual Care Group

SUMMARY:
The goal of this behavioral research study is to create and study a Mindfulness-Based Addiction Treatment (MBAT) for nicotine dependence. Mindfulness is a method to help focus attention on being in the "here and now." It can be learned through training in how to control one's attention. It is usually taught through meditation. The overarching goals of the study are to evaluate the efficacy of MBAT for nicotine dependence and the mechanisms and effects posited to mediate MBAT's impact on abstinence.

DETAILED DESCRIPTION:
This 3-group randomized clinical trial will develop and evaluate a Mindfulness-Based Addiction Treatment (MBAT) for nicotine dependence. Mindfulness reflects a purposeful control of attention and can be learned through training in attentional control procedures.

Current cigarette smokers (N=550; 400 in formal study; up to 80-150 pilot) will be randomly assigned to Usual Care (UC), Standard Treatment (ST) or MBAT. UC will be four 5-10 minute counseling sessions following the problem-solving approach in the Treating Tobacco Use and Dependence Clinical Practice Guideline (Guideline). ST is a standard smoking cessation group program using a problem-solving/coping skills approach. MBAT is a group smoking cessation program derived from Mindfulness-Based Stress Reduction (MBSR) and Mindfulness-Based Cognitive Therapy. MBAT will not alter the basic mindfulness approach used in MBCT and MBSR, but will replace depression-related material with smoking cessation strategies from the Guideline. All participants will receive nicotine patches and self-help materials. MBAT mechanisms and effects will be assessed using "implicit" cognitive psychological measures and computer-administered questionnaires. Participants will be tracked from baseline through 4 (UC) or 8 (ST and MBAT) treatment visits and follow-up visits 1 and 23 weeks post-treatment.

The overarching goals are to evaluate MBAT's efficacy for nicotine dependence and the mechanisms and effects posited to mediate MBAT's impact on abstinence.

Primary specific aims are to:

1. Examine the effects of MBAT on abstinence rates
2. Examine the effects of MBAT on mindfulness/metacognitive awareness, attentional control, smoking automaticity, smoking associations in memory, negative affect, depression, stress, affect regulation expectancies, self-efficacy, withdrawal, and coping across the pre- and post-cessation period, and whether these variables mediate MBAT effects on abstinence.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or above
2. Current smoker with a history of at least five cigarettes/day for the past year
3. Motivated to quit within the next 30 days (preparation stage)
4. Participants must provide a viable home address and a functioning home telephone number
5. Can read and write in English
6. Register "8" or more on a carbon monoxide breath test
7. Provide viable collateral contact information

Exclusion Criteria:

1. Contraindication for nicotine patch use
2. Regular use of tobacco products other than cigarettes (cigars, pipes, smokeless tobacco)
3. Use of bupropion or nicotine patch replacement products other than the study patches
4. Pregnancy or lactation
5. Another household member enrolled in the study
6. Active substance dependence (exclusive of nicotine dependence)
7. Current psychiatric disorder; current use of psychotropic medication
8. Participation in a smoking cessation program or study during the past 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2005-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David W Wetter, Ph.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Jackson S, Brown J, Norris E, Livingstone-Banks J, Hayes E, Lindson N. Mindfulness for smoking cessation. Cochrane Database Syst Rev. 2022 Apr 14;4(4):CD013696. doi: 10.1002/14651858.CD013696.pub2. PMID 35420700
- [Derived] Vidrine JI, Businelle MS, Reitzel LR, Cao Y, Cinciripini PM, Marcus MT, Li Y, Wetter DW. Coping Mediates the Association of Mindfulness with Psychological Stress, Affect, and Depression Among Smokers Preparing to Quit. Mindfulness (N Y). 2015 Jun;6(3):433-443. doi: 10.1007/s12671-014-0276-4. Epub 2014 Jan 18. PMID 28191263
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Houston metropolitan area via local print media. All data collected between January 2007 to February 2010.
Pre-assignment Details: Out of the 650 participants, 412 were on the formal clinical trial and 238 were registered under the pilot phase which were not included in the formal clinical trial and no data collected for those 238 participants.
Groups:
- Cognitive Behavioral Treatment (CBT): Standard Care Group (ST) is 6 weeks of nicotine patch therapy, a Self-help guide and In-person group therapy/counseling (8 sessions over 8 weeks) based upon Treating Tobacco Use and Dependence Clinical Practice Guideline
Period: Overall Study
Arm/Group | Usual Care Group | Cognitive Behavioral Treatment (CBT) | Mindfulness-Based Treatment Group (MBAT)
Started | 103 | 155 | 154
4-Week Follow Up | 78 | 132 | 128
26- Week Follow Up | 66 | 101 | 103
Completed | 66 | 101 | 103
Not Completed | 37 | 54 | 51
Not completed — Lost to Follow-up | 37 | 54 | 51

BASELINE CHARACTERISTICS:
Population: 238 were registered under the pilot phase which were not included in the formal clinical trial and no data collected for those 238 participants.
Groups:
- Usual Care Group (UC): 6 wks of nicotine patch therapy, self-help guide and in-person individual counseling (4 sessions in 8 weeks) based on Tobacco Use and Dependence Clinical Practice Guideline
- Cognitive Behavioral Treatment (CBT): 6 wks of nicotine patch therapy, self-help guide and in-person group counseling (8 sessions in 8 weeks) based on Treating Tobacco Use and Dependence Clinical Practice Guideline
- Mindfulness-Based Treatment Group (MBAT): 6 wks of nicotine patch therapy; self-help guide; and in-person group counseling (8 sessions in 8 weeks) using a Mindfulness-Based Addiction Treatment for nicotine dependence
- Total: Total of all reporting groups
Arm/Group | Usual Care Group (UC) | Cognitive Behavioral Treatment (CBT) | Mindfulness-Based Treatment Group (MBAT) | Total
Number analyzed (Participants) | 103 | 155 | 154 | 412
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 103 | 155 | 154 | 412
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (12.5) | 48.8 (11.9) | 48.4 (11.7) | 48.7 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 84 | 84 | 226
  Male | 45 | 71 | 70 | 186
Region of Enrollment [Number; unit: participants]
  United States | 103 | 155 | 154 | 412
Kentucky Inventory of Mindfulness Skills (KIMS) [Mean (Standard Deviation); unit: KIMS Score] — The Kentucky Inventory of Mindfulness Skills (KIMS) is a self-report inventory for the assessment of mindfulness skills (including subscales for observing (15-59), describing (10-40), acting with awareness (15-48), and accept(13-45) . Items are rated on a 5 point Likert scale ranging from 1 (never or very rarely true) to 5 (almost always or always true). Items reflect either direct descriptions of the mindfulness skills, or they describe the absence of that skill and are reverse scored. The minimum score 10 and maximum score 59. Higher-scores reflect more mindfulness.
  KIMS Score | 31.9 (4.0) | 31.9 (3.6) | 32.0 (3.8) | 32.0 (3.8)
Mindful Attention Awareness Scale (MAAS) [Mean (Standard Deviation); unit: MAAS Score] — The Mindful Attention Awareness Scale (MAAS) is a 15 item self-report questionnaire measuring mindfulness. To score the scale, simply compute a mean (average) of the 15 items. Items are rated on using the 1-6 scale ranging from 1 (almost always) to 6 (almost never). Indicates currently how frequently or infrequently each experience.
  MAAS Score | 4.2 (.9) | 4.3 (.9) | 4.3 (1.0) | 4.3 (.9)
Nicotine Dependence - Cigarettes per day [Mean (Standard Deviation); unit: Cigarettes per day] — Nicotine Dependence was assessed at baseline using the Heaviness of Smoking Index (HIS). The HSI comprises the two items from the Fagerstrom Test for Nicotine Dependence (FTND) that most strongly predict smoking relapse, cigarettes per day (CPD) and minutes to the first cigarette after waking.
  Cigarettes per day | 19.3 (8.6) | 19.9 (9.3) | 20.3 (11.7) | 19.9 (10.1)
Nicotine Dependence - Participants reported smoking their first cigarette with 5 minutes of walking [Count of Participants; unit: Participants] — Nicotine Dependence was assessed at baseline using the Heaviness of Smoking Index (HIS). The HSI comprises the two items from the Fagerstrom Test for Nicotine Dependence (FTND) that most strongly predict smoking relapse, cigarettes per day (CPD) and minutes to the first cigarette after waking.
  Participants | 39 | 61 | 59 | 159
Demographics (Education) [Count of Participants; unit: Participants] — Years of Education
  Participants
    < High School | 10 | 13 | 14 | 37
    High School/GED | 25 | 37 | 39 | 101
    Some College | 52 | 76 | 67 | 195
    4-year College Degree | 10 | 17 | 28 | 55
    > 4-year College Degree | 6 | 11 | 6 | 23
Demographics (Household Income) [Count of Participants; unit: Participants] — Income: self-reported household income
  Participants
    < $30,000/year | 61 | 89 | 87 | 237
    > $30,000/year | 42 | 66 | 67 | 175
Demographics (Spouse/Partner) [Count of Participants; unit: Participants] — Relationship status: self-report of participants with no partner
  Participants | 76 | 103 | 109 | 288
Demographics (History of Depression) [Count of Participants; unit: Participants] — The Center of Epidemiologic Studies Depression Scale (CES-D) assesses depressive symptoms in community non-clinical populations
  Participants | 22 | 27 | 22 | 71

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Smoking Abstinence
Description: Biochemically verified 7-day point prevalence abstinence rates based on a completers-only approach.
Time Frame: 4 weeks post quit day (one week following the end of treatment)
Population: Completers-only
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group (UC) | Cognitive Behavioral Treatment (CBT) | Mindfulness-Based Treatment Group (MBAT)
Number analyzed (Participants) | 66 | 101 | 103
Participants | 21 | 39 | 43

2. Primary Outcome: Smoking Abstinence
Description: Biochemically verified 7-day point prevalence abstinence rates using an intent-to-treat approach
Time Frame: 26 weeks post quit day
Population: Completers Only
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group (UC) | Cognitive Behavioral Treatment (CBT) | Mindfulness-Based Treatment Group (MBAT)
Number analyzed (Participants) | 66 | 101 | 103
Participants | 13 | 24 | 20

3. Primary Outcome: Smoking Abstinence
Description: Biochemically verified 7-day point prevalence abstinence rates using an intent-to-treat approach
Time Frame: 4 weeks post quit day (one week following the end of treatment)
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group (UC) | Cognitive Behavioral Treatment (CBT) | Mindfulness-Based Treatment Group (MBAT)
Number analyzed (Participants) | 103 | 155 | 154
Participants | 25 | 50 | 52

4. Primary Outcome: Smoking Abstinence
Description: Biochemically verified 7-day point prevalence abstinence rates using an intent-to-treat approach
Time Frame: 26 weeks post quit day
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group (UC) | Cognitive Behavioral Treatment (CBT) | Mindfulness-Based Treatment Group (MBAT)
Number analyzed (Participants) | 103 | 155 | 154
Participants | 12 | 24 | 53

ADVERSE EVENTS:
Time Frame: Adverse event data collected up to 32 weeks of treatment.
Description: MD Anderson requires that all Protocol PIs and their designees report all Serious Adverse Events.No SAE's nor Adverse Events occurred in this protocol to the MD Anderson IRB on an ongoing bases using a systematic approach with standardized forms. SAE's and AE's are reported as they occur and during each continuation report submission. 238 participants were registered under the pilot phase which were not included in the formal clinical trial and no data collected.participants.
Groups:
- Usual Care Group: Usual Care (UC) 6 weeks of nicotine patch therapy, Self-help guide & In-person individual counseling (4 sessions over 8 weeks)
- Standard Care Group: Standard Care Group (ST) 6 weeks of nicotine patch therapy, Self-help guide & In-person group therapy/counseling (8 sessions over 8 weeks)
- Mindfulness-Based Treatment Group (MBAT): MBAT 6 weeks of nicotine patch therapy; Self-help guide; & In-person group therapy/counseling (8 sessions over 8 weeks) using a MBAT for nicotine dependence.
Arm/Group | Usual Care Group | Standard Care Group | Mindfulness-Based Treatment Group (MBAT)
Serious Adverse Events (participants affected / at risk) | 0/103 | 0/155 | 0/154
Other Adverse Events (participants affected / at risk) | 0/103 | 0/155 | 0/154

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes